CLINICAL TRIAL: NCT01053728
Title: Randomized, Double-blind, Euglycemic Glucose Clamp Study of Four Formulations of SAR161271, in Single Doses in Healthy Subjects and Single Ascending Doses in Patients With Type 1 Diabetes Mellitus
Brief Title: Study of How Single Rising Doses of SAR161271 Are Absorbed and Act in Patients With Type 1 Diabetes Mellitus (T1DM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TDU10987; TDU10948
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 : SAR161271 0.3 U/kg (Experimental): Cross-over design of four formulation of SAR161271 0.3U/kg or insulin glargine administered as a single dose in the morning between about 11h00 and about 12h00; fasting for about 12h before and for the duration of the clamp
  Interventions: Drug: SAR161271; Drug: Insulin glargine HOE901
- Cohort 2 : SAR161271 0.6 U/kg (Experimental): Cross-over design of four formulation of SAR161271 0.6U/kg or insulin glargine administered as a single dose in the morning between about 11h00 and about 12h00; fasting for about 12h before and for the duration of the clamp
  Interventions: Drug: SAR161271; Drug: Insulin glargine HOE901
- Cohort 3 : SAR161271 1.2 U/kg (Experimental): Cross-over design of four formulation of SAR161271 1.2 U/kg or insulin glargine administered as a single dose in the morning between about 11h00 and about 12h00; fasting for about 12h before and for the duration of the clamp
  Interventions: Drug: SAR161271; Drug: Insulin glargine HOE901

INTERVENTIONS:
Drug: SAR161271 — Pharmaceutical form:Solution for injection
  Route of administration: subcutaneous
Drug: Insulin glargine HOE901 — Pharmaceutical form:Solution for injection
  Route of administration: subcutaneous

SUMMARY:
Primary Objective:

- To establish initial safety/tolerability and pharmacodynamic and pharmacokinetic profiles of four formulations of SAR161271 in patients with T1DM.

Secondary Objective:

- To establish relative potency of SAR161271 compared with insulin glargine in patients with T1DM

DETAILED DESCRIPTION:
The total per patient is between 31 and 67 days; including post-study visit between 108 and 172 days. In case of an additional late post-study visit after last dosing, approximately 213 to 279 days, broken down as follows:

* Screening: 3 to 27 days;
* Treatment Periods each 1 day with institutionalisation from Day -1 to Day 3;
* Wash-out between doses: 7 to 10 days;
* End of Study visit: 7 to 10 days after last dose.
* Post-study visit 84 to 112 days after last dosing. If necessary, additional post-study visit 6 to 7 months after last dosing.

ELIGIBILITY:
Inclusion criteria:

* Patients who have type 1 diabetes mellitus (T1DM) as defined by American Diabetes Association average total insulin dose of <1.2 U/kg/day
* Fasting negative serum C-peptide (<0.3 nmol/L)
* Glycated hemoglobin (HbA1c) < or = 9%
* Stable insulin regimen for at least 2 months before the study
* Body weight between 50-110 kg inclusive; body mass index between 18-30 kg/m2, inclusive
* Certified as healthy for T1DM by a comprehensive clinical assessment

Exclusion criteria:

* Any history or presence of clinically relevant (for T1DM) cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness, or major diabetic complications such as diabetic retinopathy.
* Blood donation, any volume, within 1 month before inclusion.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician
* Regular use of any medication other than insulins in the last month before study start with the exception of thyroid hormones, metformin, lipid-lowering and antihypertensive drugs
* Positive reaction to any of the following tests: hepatitis B surface (HBs) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus (HIV) 1 antibodies, anti-HIV2 antibodies.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
- Safety in terms of adverse and serious adverse events, vital signs, ECG, safety laboratory for each cohort | up to 7 days after dose
- Pharmacodynamics (Glucose infusion rate) time-action profile | up to 30 hours after dose

SECONDARY OUTCOMES:
- Pharmacokinetic parameters | up to 168 hours after dose
- anti-insulin antibody production | pre-dose and after 4th dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Berlin, Germany